CLINICAL TRIAL: NCT00985946
Title: A Phase II Trial of Panobinostat in Patients With Neuroendocrine Tumors
Brief Title: Study of Panobinostat in Patients With Neuroendocrine Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study did not meet statistical requirements to continue.
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO08209; CLBH589BUS38T (Other Grant/Funding Number: Novartis); 2010-0050 (Other: Institutional Review Board); 2014-1298 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); NCI-2011-00320 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2009-09-25; First posted 2009-09-29 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2017-06

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- panobinostat (Experimental): This is a single arm trial. All patients will take panobinostat
  Interventions: Drug: panobinostat (LBH589)

INTERVENTIONS:
Drug: panobinostat (LBH589) — Panobinostat will be taken once daily at 20 mg three times a week (every Monday, Wednesday, Friday). It will be taken as long as patients are benefiting from treatment.

SUMMARY:
This summary will use Panobinostat (LBH589) in patients with neuroendocrine tumors to see how the patient's tumor responds to panobinostat. Additionally, this study will examine how long it takes neuroendocrine tumor patient's cancer to progress while taking the drug and examine the overall survival of patients using panobinostat. Also, the study will examine the toxicity and tolerability of panobinostat in the patient population. Finally, this study will look at the effect of panobinostat on Notch 1 signaling before and after treatment with panobinostat.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, metastatic, low grade neuroendocrine neoplasms. Small cell lung cancers, paragangliomas, and pheochromocytomas are excluded
* Must have measurable disease as defined by RECIST
* 4 weeks from completion of major surgery, chemotherapy, or other systemic therapy or local liver therapy to study registration. Concurrent octreotide is allowed.
* Not allowed to be on concurrent chemotherapy or radiation
* 18 years of age or older
* ECOG Performance status of equal to or less than 2
* Able to sign and date a written informed consent prior to participation in the study
* Baseline MUGA or ECHO must demonstrate LVEF greater than or equal to the lower limit of the institutional normal
* Must have the following laboratory criteria: Neutrophil count greater than 1500/mm3, platelet count greater than 100,000/mm3L, hemoglobin greater than or equal to 9 g/dL, AST/SGOT and ALT/SGPT less than or equal to 2.5 x ULN, serum bilirubin less than or equal to 1.5 x ULN, serum creatinine less than or equal to 1.5 x ULN, total serum calcium greater than or equal to LLN, serum potassium greater than or equal to LLN, serum sodium greater than or equal to LLN, serum albumin greater than or equal to LLN or 3g/dl,
* Women of child bearing potential must have a negative urine pregnancy test within 72 hours of first administration of study treatment and must be willing to use two methods of contraception
* Patients with a history of hypertension must be well controlled (to less than 150/90 mmHg) on a stable regimen of anti-hypertensive therapy

Exclusion Criteria:

* Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer
* Patients who will need valproic acid for any medical condition during the study or within 5 days prior to the first panobinostat treatment
* Impaired cardiac function including any of the following: Screening ECG with a QTc greater than 450 msec, patients with congenital long QT syndrome, history of unsustained ventricular tachycardia, any history of ventricular fibrillation or torsades de pointes, bradycardia defined as heart rate less than 50 beats per minutes, patients with a myocardial infarction or unstable angina within 6 months of study entry, congestive heart failure, right bundle branch block or left anterior hemiblock
* Uncontrolled hypertension
* Unresolved diarrhea greater than CTCAE grade 1
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral panobinostat
* Other concurrent sever and/or uncontrolled medical conditions
* Patients with a history of another primary malignancy that, in the opinion of the investigator, would interfere with the assessment of the primary endpoint of the study
* Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis C, baseline testing is not required
* Any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent
* Any medication which may cause QTc prolongation or inducing torsades de pointes
* Use of concomitant medications that may interact with panobinostat

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noelle LoConte, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Jin N, Lubner SJ, Mulkerin DL, Rajguru S, Carmichael L, Chen H, Holen KD, LoConte NK. A Phase II Trial of a Histone Deacetylase Inhibitor Panobinostat in Patients With Low-Grade Neuroendocrine Tumors. Oncologist. 2016 Jul;21(7):785-6. doi: 10.1634/theoncologist.2016-0060. Epub 2016 Jun 3. PMID 27261467
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study actively recruited from April 2010 through May 2011 at a large cancer center in Wisconsin.
Groups:
- Panobinostat: Adult patients with histologically confirmed, metastatic, low-grade NETs and an Eastern Cooperative Oncology Group (ECOG) performance status of ≤2 were treated with oral panobinostat 20 mg once daily three times per week. Treatment was continued until patients experienced unacceptable toxicities or disease progression. The study was stopped at planned interim analysis based on a Simon two-stage design.
Period: Overall Study
Arm/Group | Panobinostat
Started | 15 (Eighty-seven percent (n=13) were evaluable for response.)
Completed | 8
Not Completed | 7
Not completed — Lost to Follow-up | 6
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Panobinostat
Number analyzed (Participants) | 15
Age, Customized [Number; unit: participants]
  40-49 years of age | 3
  50-59 years of age | 5
  60-69 years of age | 4
  70-79 years of age | 2
  >= 80 years of age | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate of Patients With Gastrointestinal Neuroendocrine Tumors Using Response Evaluation Criteria in Solid Tumors (RECIST) Criteria.
Description: Confirmed anti-tumor response rate will be validated by the Response Evaluation Criteria in Solid Tumors (RECIST). All participants included in the study will be assessed for response to the proposed panobinostat treatment, even if there are protocol treatment deviations. Each participant will be assigned one of the following categories: complete response, partial response, stable disease, progressive disease, early death from malignant disease, early death from toxicity, early death because of other cause, or unknown.
Time Frame: every 8 weeks, up to 5 years
Measure: Number; unit: participants
Arm/Group | Panobinostat
Number analyzed (Participants) | 15
participants
  Stable Disease | 15
  Complete Response | 0
  Partial Response | 0
  Progressive Disease | 0
  Early death from malignant disease | 0
  Early death from toxicity | 0
  Early death because of other cause | 0
  Unknown | 0

2. Secondary Outcome: Number of Participants With Toxicities
Description: Evaluate the toxicity and tolerability of panobinostat in the patient population
Time Frame: up to 5 years
Measure: Number; unit: participants
Arm/Group | Panobinostat
Number analyzed (Participants) | 15
participants | 5

3. Secondary Outcome: Evaluate the Time to Progression for Patients With Gastrointestinal Neuroendocrine Tumors Treated With Panobinostat
Time Frame: Up to 5 years
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Panobinostat
Number analyzed (Participants) | 15
months | 9.9 [4.1 to 16.9]

4. Secondary Outcome: Delineate the Expression of Notch 1 in Neuroendocrine Tumor Samples Before and During Treatment With Panobinostat
Description: The expression of Notch 1 in neuroendocrine tumor samples will be evaluated prior to Cycle 1 Day 1 dose and at the end of Cycle 2 of treatment of treatment.
Time Frame: Pre-treatment and up to week 12
Population: Data to delineate the expression of Notch 1 in neuroendocrine tumor samples was not collected. The question regarding the role of Notch1 in well-differentiated NET remains unanswered.
Arm/Group | Panobinostat
Number analyzed (Participants) | 0

5. Secondary Outcome: Evaluate the Overall Survival of Patients With Gastrointestinal Neuroendocrine Tumors Treated With Panobinostat
Time Frame: Up to 5 years
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Panobinostat
Number analyzed (Participants) | 15
months | 47.27 [17.87 to NA] — Not reached.

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 5 years.
Description: Grade refers to the severity of the Adverse Event (AE) from grades 1 through 5, where 1 is a mild AE, and 5 is death related to an adverse AE.
  Systematic Adverse Event assessment included regular assessment of subjects by the treating investigator, including physical exam, ECOG performance status, ECG, and lab assessments.
Groups:
- Panobinostat: Adult patients with histologically confirmed, metastatic, low-grade NETs and an Eastern Cooperative Oncology Group (ECOG) performance status of ≤2 were treated with oral panobinostat 20 mg once daily three times per week. Treatment was continued until patients experienced unacceptable toxicities or disease progression. The study was stopped at planned interim analysis based on a Simon two-stage design. Fifteen patients were accrued, and 13 were evaluable for response. No responses were seen, but the stable disease rate was 100%. The median progression-free survival (PFS) was 9.9 months, and the median overall survival was 47.3 months. Fatigue (27%), thrombocytopenia (20%), diarrhea (13%), and nausea (13%) were the most common related grade 3 toxicities. There was one grade 4 thrombocytopenia (7%). These results did not meet the prespecified criteria to open the study to full accrual.
Arm/Group | Panobinostat
Serious Adverse Events (participants affected / at risk) | 6/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panobinostat (N=15)
Grade 3 albumin, serum low (Metabolism and nutrition disorders) | 1 (1)
Grade 1 creatinine (Metabolism and nutrition disorders) | 1 (1)
Grade 3 diarrhea (Gastrointestinal disorders) | 2 (2)
Grade 3 febrile neutropenia (Infections and infestations) | 1 (1)
Grade 1 glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1)
Grade 2 hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Grade 3 hypotension (Cardiac disorders) | 1 (1)
Grade 5 hypotension (death) (Cardiac disorders) | 1 (1) — Subject expired less than 30 days off study
Grade 3 infection (Infections and infestations) | 1 (1)
Grade 3 lipase (Metabolism and nutrition disorders) | 1 (1)
Grade 4 lipase (Metabolism and nutrition disorders) | 1 (1)
Grade 1 magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Grade 3 pain (General disorders) | 2 (2)
Grade 4 pain (General disorders) | 1 (1)
Grade 2 pancreatitis (Hepatobiliary disorders) | 1 (1)
Grade 4 platelets (thrombocytopenia) (Blood and lymphatic system disorders) | 1 (1)
Grade 3 Pneumotosis Coli (Gastrointestinal disorders) | 1 (1)
Grade 1 potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Grade 3 small bowel NOS (Gastrointestinal disorders) | 1 (1)
Grade 1 sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panobinostat (N=15)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 8 (27)
Alkaline phosphatase (Investigations) | 8 (15)
Allergic rhinitis (Immune system disorders) | 1 (1)
Allergy/Immunology (Immune system disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 6 (18)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 1 (1)
Auditory/Ear (Ear and labyrinth disorders) | 1 (1)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 3 (6)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (4)
Cervical spine-range of motion (Musculoskeletal and connective tissue disorders) | 1 (1)
Cholesterol, serum-high (hypercholesteremia) (Investigations) | 5 (26)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine (Investigations) | 8 (43)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 13 (52)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Edema: limb (Blood and lymphatic system disorders) | 2 (3)
Elevated Triglycerides (Metabolism and nutrition disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 15 (68)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 4 (9)
Flushing (Vascular disorders) | 5 (20)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 (2)
Gastrointestinal (Gastrointestinal disorders) | 3 (3)
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 8 (21)
Gingivitis (Infections and infestations) | 1 (1)
Glomerular filtration rate (Renal and urinary disorders) | 5 (12)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 13 (61)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 2 (2)
Hemoglobin (Investigations) | 10 (42)
Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (3)
Hypotension (Vascular disorders) | 3 (5)
Infection (Infections and infestations) | 2 (3)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 2 (9)
Joint-function (Musculoskeletal and connective tissue disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 3 (18)
Lipase (Investigations) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 3 (8)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 4 (8)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 3 (3)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 2 (3)
Musculoskeletal/Soft Tissue (Musculoskeletal and connective tissue disorders) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 13 (39)
Neuropathy: sensory (Nervous system disorders) | 2 (8)
Neutrophils/granulocytes (ANC/AGC) (Nervous system disorders) | 4 (16)
Pain (General disorders) | 11 (40)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (8)
Platelets (Blood and lymphatic system disorders) | 13 (73)
Potassium, serum-high (hyperkalemia) (Investigations) | 3 (9)
Potassium, serum-low (hypokalemia) (Investigations) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 5 (18)
Sweating (diaphoresis) (General disorders) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 4 (5)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1)
Thyroid function, high (hyperthyroidism, thyrotoxicosis) (Endocrine disorders) | 4 (6)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 8 (26)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (4)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 8 (51)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (17)
Weight loss (Investigations) | 9 (37)

LIMITATIONS AND CAVEATS:
This study was terminated early because of the use of objective response rate as the primary outcome measure, which is a shortcoming of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No